CLINICAL TRIAL: NCT03268382
Title: PiSARRO-R: p53 Suppressor Activation in Platinum-Resistant High Grade Serous Ovarian Cancer, a Phase II Study of Systemic Pegylated Liposomal Doxorubicin Chemotherapy With APR-246
Brief Title: p53 Activation in Platinum-Resistant High Grade Serous Ovarian Cancer, a Study of PLD With APR-246
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aprea Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APR-486
Record Dates: First submitted 2017-08-24; First posted 2017-08-31 (Actual); Results first posted 2022-07-21 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: High-grade Serous Ovarian Cancer
Keywords: Ovarian Cancer; Ovarian Carcinoma; High Grade Serous Ovarian Cancer; Recurrent Cancer; Resistant Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Recurrence | interventions — eprenetapopt

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- APR-246 + PLD (Experimental)
  Interventions: Drug: APR-246; Drug: Pegylated Liposomal Doxorubicin Hydrochloride (PLD)

INTERVENTIONS:
Drug: APR-246 — Intravenous infusion
Drug: Pegylated Liposomal Doxorubicin Hydrochloride (PLD) — Intravenous infusion

SUMMARY:
The purpose of this study is to make a preliminary assessment of the efficacy of a combined APR-246 and PLD chemotherapy regimen in patients with platinum-resistant recurrent high grade serous ovarian cancer (HGSOC) with mutated TP53. In addition, the study aims to assess the safety profile of the combined APR-246 and PLD chemotherapy regimen, to evaluate potential biomarkers, and to assess the biological activity in tumor and surrogate tissues. The trial will enroll at least 25 evaluable patients.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed High Grade Serous Ovarian Cancer, and positive nuclear immunohistochemical (IHC) staining for p53
* Disease Progression between 4 weeks - 6 months after the last platinum-based treatment was administered
* At least a single measurable lesion
* Adequate organ function prior to registration
* Toxicities from previous cancer therapies (excluding alopecia) must have recovered to grade 1 (defined by National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] version 4.0). Chronic stable grade 2 peripheral neuropathy secondary to neurotoxicity from prior therapies may be considered on a case by case basis
* ECOG performance status of 0 to 2

Exclusion Criteria:

* Prior exposure to cumulative doses of doxorubicin >400 mg/m2 or epirubicin >720 mg/m2
* Hypersensitivity to PLD or to any of the excipients
* Unable to undergo imaging by either CT scan or MRI
* Evidence of any other medical conditions (such as psychiatric illness, infectious diseases, neurological conditions, physical examination or laboratory findings) that may interfere with the planned treatment, affect patient compliance or place the patient at high risk from treatment related complications
* Concurrent malignancy requiring therapy (excluding non-invasive carcinoma or carcinoma in situ)
* Is taking concurrent (or within 4 weeks prior to registration) chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy that is considered to be investigational (i.e., used for non-approved indications(s) and in the context of a research investigation). Supportive care measures are allowed. Palliative limited radiation therapy for pain reduction is allowed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2019-07-10 (Actual); Study Completion 2019-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charlie Gourley, BSc, MB ChB, PhD, FRCP, Principal Investigator — Edinburgh Cancer Research Centre, The University of Edinburgh
Locations (12):
- Belgium (3):
  - Medische oncologie, Universitair Ziekenhuis Gent, Ghent
  - Leuven University Hospitals, Leuven
  - Centre Hospitalier Universitaire de Liège, Liège
- Spain (5):
  - Institut Català d'Oncologia, Hospital Germans Trias i Pujol, Badalona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Clinico Universitario de Valencia, Valencia
- United Kingdom (4):
  - Cambridge Cancer Trials Centre, Cambridge University Hospitals NHS Foundation Trust, Addenbrooke's Hospital, Cambridge
  - Edinburgh Cancer Research Centre, The University of Edinburgh, Edinburgh
  - The Royal Marsden NHS Foundation Trust, London
  - Imperial College London, Hammersmith Hospital Campus, London

REFERENCES:
- [Background] Lehmann S, Bykov VJ, Ali D, Andren O, Cherif H, Tidefelt U, Uggla B, Yachnin J, Juliusson G, Moshfegh A, Paul C, Wiman KG, Andersson PO. Targeting p53 in vivo: a first-in-human study with p53-targeting compound APR-246 in refractory hematologic malignancies and prostate cancer. J Clin Oncol. 2012 Oct 10;30(29):3633-9. doi: 10.1200/JCO.2011.40.7783. Epub 2012 Sep 10. PMID 22965953
- [Background] Deneberg S, Cherif H, Lazarevic V, Andersson PO, von Euler M, Juliusson G, Lehmann S. An open-label phase I dose-finding study of APR-246 in hematological malignancies. Blood Cancer J. 2016 Jul 15;6(7):e447. doi: 10.1038/bcj.2016.60. No abstract available. PMID 27421096
- See also: Aprea Therapeutics AB's website (Sponsor) — http://www.aprea.com

RESULTS

PARTICIPANT FLOW:
Groups:
- APR-246 (4.5g/6hr) + PLD; APR-246 (4.5g/3hr) +PLD; APR-246 (4.5g/4hr) +PLD; APR-246 (3.7g/4hr) +PLD: APR-246: Intravenous infusion Pegylated Liposomal Doxorubicin Hydrochloride (PLD): Intravenous infusion
Period: Overall Study
Arm/Group | APR-246 (4.5g/6hr) + PLD | APR-246 (4.5g/3hr) +PLD | APR-246 (4.5g/4hr) +PLD | APR-246 (3.7g/4hr) +PLD
Started | 28 | 3 | 2 | 3
Completed | 28 | 3 | 2 | 3
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients with Pt-resistant HGSOC with TP53 mutation.
Groups:
- APR-246 (4.5g/3hr) + PLD; APR-246 (4.5g/4hr) + PLD; APR-246 (3.7g/4hr) + PLD: APR-246: Intravenous infusion Pegylated Liposomal Doxorubicin Hydrochloride (PLD): Intravenous infusion
- Total: Total of all reporting groups
Arm/Group | APR-246 (4.5g/6hr) + PLD | APR-246 (4.5g/3hr) + PLD | APR-246 (4.5g/4hr) + PLD | APR-246 (3.7g/4hr) + PLD | Total
Number analyzed (Participants) | 28 | 3 | 2 | 3 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 21 | 2 | 1 | 2 | 26
  >=65 years | 7 | 1 | 1 | 1 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 3 | 2 | 3 | 36
  Male | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 27 | 3 | 2 | 3 | 35
  Asian | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Belgium | 4 | 0 | 0 | 0 | 4
  United Kingdom | 3 | 3 | 2 | 3 | 11
  Spain | 21 | 0 | 0 | 0 | 21

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 18 months
Population: A total of 36 patients were enrolled in this Phase II study. Of the 36 patients, 28 patients were in the main study, 4.5g/6hr dose cohort; 8 patients were in the sub-study as follows: 3 patients were in the 4.5g/3hr dose cohort; 2 patients were in the 4.5g/4hr dose cohort and 3 patients were in the 3.7g/4hr dose cohort.
  The 23 Efficacy Evaluable Patients from the Main Study (APR-246 (4.5g/6hr) + PLD) are part of the analysis reported below.
Measure: Count of Participants; unit: Participants
Arm/Group | APR-246 (4.5g/6hr) + PLD | APR-246 (4.5g/3hr) + PLD | APR-246 (4.5g/4hr) + PLD | APR-246 (3.7g/4hr) + PLD
Number analyzed (Participants) | 23 | 3 | 2 | 3
Participants
  Partial Response (PR) | 1 | 0 | 0 | 0
  Stable Disease (SD) | 15 | 2 | 1 | 1
  Progressive Disease (PD) | 7 | 0 | 1 | 2
  Not Evaluable | 0 | 1 | 0 | 0
  Disease Control Rate (CR+PR+SD) | 16 | 0 | 0 | 0

2. Secondary Outcome: Treatment-emergent Adverse Events With Combined APR-246 and PLD Regimen
Description: Treatment emergent adverse events (TEAEs) were defined as AEs that occurred on or after the first dose of study medication up to and including 30 days after last dose. AEs were graded according to NCI CTCAE (Version 4.0). Patients with multiple TEAEs were only counted once within a summary category: SOC, PT, maximum grade, or relationship to treatment. Patients with events in more than one category were counted once within each category.
Time Frame: Treatment emergent adverse events (TEAEs) were defined as AEs that occurred on or after the first dose of study medication up to and including 30 days after last dose. Median number of 28d Cycles=2.5 (Min = 1, Max = 14)
Measure: Count of Participants; unit: Participants
Arm/Group | APR-246 (4.5g/6hr) + PLD | APR-246 (4.5g/3hr) + PLD | APR-246 (4.5g/4hr) + PLD | APR-246 (3.7g/4hr) + PLD
Number analyzed (Participants) | 28 | 3 | 2 | 3
Participants
  With Any Treatment-Emergent Adverse Events (TEAEs) | 28 | 3 | 2 | 3
  With APR-246 Related TEAEs | 25 | 3 | 2 | 3
  With PLD Related TEAEs | 24 | 3 | 2 | 3
  With Severity Grade >=3 | 14 | 3 | 2 | 3
  With Severity Grade >=3 APR-246 Related TEAEs | 6 | 2 | 2 | 2
  With Severity Grade >=3 PLD Related TEAEs | 7 | 2 | 0 | 2
  With Any Serious AEs | 11 | 1 | 1 | 2
  With Any Serious, APR-246 Related AEs | 4 | 1 | 1 | 1
  With Any Serious, PLD Related AEs | 2 | 1 | 0 | 1
  Who Discontinued APR-246 Due to TEAEs | 2 | 1 | 0 | 0
  Who Discontinued PLD Due to TEAEs | 0 | 0 | 0 | 0
  Who Died Due to any TEAEs | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events (TEAEs) were defined as AEs that occurred on or after the first dose of study medication up to and including 30 days after last dose. Median number of 28d Cycles=2.5 (Min = 1, Max = 14)
Description: AEs were graded according to NCI CTCAE (Version 4.0).
Arm/Group | APR-246 (4.5g/6hr) + PLD | APR-246 (4.5g/3hr) + PLD | APR-246 (4.5g/4hr) + PLD | APR-246 (3.7g/4hr) + PLD
All-Cause Mortality (participants affected / at risk) | 9/28 | 1/3 | 0/2 | 1/3
Serious Adverse Events (participants affected / at risk) | 11/28 | 1/3 | 1/2 | 2/3
Other Adverse Events (participants affected / at risk) | 28/28 | 3/3 | 2/2 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | APR-246 (4.5g/6hr) + PLD (N=28) | APR-246 (4.5g/3hr) + PLD (N=3) | APR-246 (4.5g/4hr) + PLD (N=2) | APR-246 (3.7g/4hr) + PLD (N=3)
Intestinal obstruction (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peritoneal fibrosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (6) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | APR-246 (4.5g/6hr) + PLD (N=28) | APR-246 (4.5g/3hr) + PLD (N=3) | APR-246 (4.5g/4hr) + PLD (N=2) | APR-246 (3.7g/4hr) + PLD (N=3)
Nausea (Gastrointestinal disorders) | 17 | 2 | 1 | 3
Vomiting (Gastrointestinal disorders) | 12 | 2 | 2 | 3
Constipation (Gastrointestinal disorders) | 11 | 1 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 9 | 0 | 1 | 3
Diarrhea (Gastrointestinal disorders) | 6 | 0 | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 3 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 6 | 3 | 1 | 3
Asthenia (General disorders) | 10 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 7 | 1 | 0 | 1
Edema peripheral (General disorders) | 4 | 1 | 0 | 0
Gait disturbance (General disorders) | 2 | 1 | 0 | 0
Device occlusion (General disorders) | 0 | 0 | 0 | 2
Infusion site vesicles (General disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 5 | 1 | 2 | 1
Dysgeusia (Nervous system disorders) | 3 | 1 | 0 | 1
Ataxia (Nervous system disorders) | 2 | 0 | 1 | 0
Dyskinesia (Nervous system disorders) | 1 | 1 | 0 | 1
Headache (Nervous system disorders) | 2 | 0 | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 1 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 1
Tremor (Nervous system disorders) | 0 | 2 | 0 | 0
Akathisia (Nervous system disorders) | 0 | 0 | 1 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 1 | 0
Apraxia (Nervous system disorders) | 0 | 0 | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 1 | 0
Nystagmus (Nervous system disorders) | 0 | 0 | 1 | 0
Paresthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0
Anemia (Blood and lymphatic system disorders) | 6 | 1 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 4 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 7 | 1 | 1 | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hypophosphatemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 3 | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 2 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 1 | 0 | 1
Device related infection (Infections and infestations) | 0 | 0 | 0 | 1
Lip infection (Infections and infestations) | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 1 | 1 | 1
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 1
Nightmare (Psychiatric disorders) | 0 | 1 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 1
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Glomerular filtration rate decreased (Investigations) | 0 | 0 | 0 | 1
Vascular disorders (Vascular disorders) | 3 | 0 | 0 | 0
Ear and labyrinth disorders (Ear and labyrinth disorders) | 1 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 1 | 0 | 0
Blepharitis (Eye disorders) | 0 | 0 | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-12): https://cdn.clinicaltrials.gov/large-docs/82/NCT03268382/Prot_SAP_000.pdf